CLINICAL TRIAL: NCT02926313
Title: The Effectiveness of Specialist Seating Provision for Nursing Home Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Seating Matters Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12/0084
Record Dates: First submitted 2016-10-03; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Physical Disability
Keywords: RCT; Specialized seating; Pressure ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Existing Seating conditions (No Intervention): This group of participants received the standard care - they continue to sit in the seating system (chair and cushion) as provided by the nursing home facility staff; selected from whatever seats the facility had available.
- Individualized Seating provision (Experimental): This group of participants were provided with a seating system that was specifically configured to match their individual postural care needs.
  Interventions: Other: Individualized Seating provision

INTERVENTIONS:
Other: Individualized Seating provision — Seating system selected and adjusted to meet individual needs.
  Arms: Individualized Seating provision

SUMMARY:
A randomized control study aimed to investigate if suitable individualized seating provision is effective for adult nursing home residents in reducing the incidence of pressure ulcers, and increasing their quality of life and functioning.

DETAILED DESCRIPTION:
The United Kingdom (UK) population demographics confirm that older people are considered to be the fastest-growing group in the population (Dunnell, 2008). In 2007, 9.8 million people were aged over 65; however, by 2032 this figure is projected to rise to 16.1 million (Dunnell, 2008). Many of these older adults will have complex health and social care needs sometimes requiring nursing home care. A high standard and quality of care within our nursing homes is essential, to be able to deal with this growing population safely and to the highest standard possible, including the provision of individualised seating assessment, prescription and provision. An individually prescribed seating system should be based upon the assessment of the person's abilities and needs, and should best position and support them for comfort and function.

When seating is not clinically suitable for the user there are many physiological and psychological implications for the user. For example, often pressure ulcers may develop. Pressure ulcers are currently a major concern for the NHS due to their prevalence, the cost of treatments and the impact on the person. Pressure ulcers can often be related to poor seating and indeed good seating can contribute to prevention and contribute to healing (Anton, 2005). Current expenditure by the NHS in the UK on pressure sores is £2.1bn annually. This equates to approximately £10,500 per sore (Bennett et al, 2004). Anecdotal evidence suggests that correct seating provision could be instrumental in depleting this cost by preventing pressure ulcers through investment in chairs before ulcers develop. This project set out to explore this topic via empirical research methods.

Research Question To identify the importance of individualised seating in reducing postural difficulties for adult residents in nursing homes.

Methods A pragmatic RCT design with qualitative and quantitative tools was used. These included: pulse oximeter readings of oxygen saturation levels and pulse rate; Braden scale of pressure risk; caregiver questionnaire; digital photographs of seated posture; and demographic information.

Participants Forty residents were recruited from three nursing homes in N.Ireland, and were randomly assigned to either the control group (continue to use existing chair) or the intervention group (use an individually configured seating system) for the 12- week trial period. At the end of the 12- week trial period there were 18 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* Adult living in one of the three nursing home facilities

Exclusion Criteria:

* Determined to be at a high risk of developing pressure ulcers (as per Braden Scale assessment)

Ages: 44 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in the Braden Scale | Change in pressure injury risk from baseline at 12 weeks
  Measures the risk of developing pressure injuries/ ulcers
Change in Oxygen saturation levels | Change in SpO2 levels from baseline at 12 weeks
  Pulse oximeter used to measure saturated oxygen levels
Seating assessment | baseline
  This measures the individual's level of sitting skills and abilities

SECONDARY OUTCOMES:
Change in sitting presentation - digitally captured | Change in sitting presentation from baseline to 12 weeks
  Visually record presentation of the resident in the seating system using digital photographs
Change in Quality of life factors - questionnaire | Change in quality of life from baseline to 12 weeks
  This questionnaire gathered perspective on changes; for example, how many times the resident needs to be moved and handled, repositioned int heir chair, whether they can feed themselves, call out to others and presence of any skin redness or skin breakdown

IPD SHARING:
Plan to Share IPD: No